CLINICAL TRIAL: NCT04032808
Title: Evaluation of the Performance of Self-monitoring Optimized by Therapeutic Education in the Recurrence of Wet Age-related Macular Degeneration (AMD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00293-54
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Monocentric and prospective study, evaluating the benefit of self-monitoring optimized by therapeutic education either by the environmental Amsler or the Amsler grid according to the patient's choice and to determine the patient's ability to determine the reality itself recidivism and therefore the need for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to a social security scheme
* Patient agreeing to participate in the process of therapeutic education.
* Centrofoveal fixation with visual acuity> 2/10
* Antecedent of at least one recurrence so that the patient is aware of the notion of recurrent chronic disease
* Intravitreal injection antecedent less than 6 months ago

Exclusion Criteria:

* Vulnerable people
* Majors subject to legal protection or unable to express their consent
* Arterial emboli disorders of less than three months such as myocardial infarction, stroke

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AMD who have had at least one recurrence after a shared education assessment in which they have indicated the need or desire to participate in the control of their disease and who agree to participate in a therapeutic education program at the Beau Soleil Clinic
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of self-monitoring by the environmental Amsler or the clinical Amsler grid according to the choice of the patient after therapeutic education. | Through study completion, on average of 1 year
  Sensitivity and specificity of self-monitoring by the environmental Amsler or the clinical Amsler grid according to the choice of the patient after therapeutic education.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Beau Soleil, Montpellier, France